CLINICAL TRIAL: NCT00119925
Title: Cost Effectiveness of Two Different Strategies to Implement the NVOG Guideline Programme on Subfertility
Brief Title: 'SPRING'-Study: "Subfertility Guidelines: Patient Related Implementation in the Netherlands Among Gynaecologists"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: J.A.M. Kremer, dept. of Obstetrics and Gynecology
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SPRING 2005-01; ZonMw grant no. 945-14-116
Record Dates: First submitted 2005-07-05; First posted 2005-07-14 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Male Infertility; Female Infertility; Ovarian Hyperstimulation Syndrome; Premature Ovarian Failure; Endometriosis
Keywords: infertility; guideline; health care implementation; intervention; gynecology
MeSH Terms: conditions — Infertility, Male; Infertility, Female; Ovarian Hyperstimulation Syndrome; Primary Ovarian Insufficiency; Endometriosis; Infertility | interventions — Patient Education as Topic; Guideline Adherence

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- minimal intervention (Active Comparator): professional audit and feedback on current practice
  Interventions: Behavioral: professional audit and feedback (guideline adherence)
- maximal intervention (Active Comparator): multi-faceted intervention consisting of professional and patient elements
  Interventions: Behavioral: patient education; Behavioral: professional audit and feedback (guideline adherence); Behavioral: professional education (communication/shared decision making); Other: information tools

INTERVENTIONS:
Behavioral: patient education — patient leaflets about national guideline contents
  Arms: maximal intervention
Behavioral: professional audit and feedback (guideline adherence) — feedback on current practice according to quality indicators
Behavioral: professional education (communication/shared decision making) — educational tools for professionals concerning communication and shared decision making
  Arms: maximal intervention
Other: information tools — tools and checklists to improve information provision
  Arms: maximal intervention

SUMMARY:
The purpose of this study is to compare two different strategies to implement the existing Guideline programme on Subfertility, as issued by the Dutch Society of Obstetrics and Gynaecology (NVOG). Therefore, an innovative patient-directed strategy will be compared to a control strategy and effectiveness, costs and feasibility of both strategies will be assessed.

DETAILED DESCRIPTION:
The Dutch Society of Obstetrics and Gynaecology (NVOG) has developed a guideline programme on Subfertility, including 9 guidelines concerning diagnosis and treatment of subfertility and a national IVF protocol.

However, guidelines in general do not implement themselves; large gaps consists between best evidence (as described in the guidelines) and practice, resulting in a large variation between professionals.

Our study will compare an innovative patient-directed strategy with a (minimal intervention) control strategy, and effectiveness, costs and feasibility of both will be assessed. We eventually aim at the most cost-effective strategy to implement the existing subfertility guideline programme.

Please Note: In our protocol, we consider only 'couples' undergoing fertility treatment; therefore, we aim at gathering information from approximately 5200 records, of both male and female participants. When reporting eventually on their treatment, we will consider them only as couples, resulting in reported numbers of approximately 2600 participating couples.

ELIGIBILITY:
Inclusion Criteria:

* each patient, male or female, visiting the OPD for a subfertility related problem or treatment
* each patient admitted to the hospital with complications of an infertility treatment

Exclusion Criteria:

* patients receiving insemination with donor sperm
* patients receiving ICSI treatment
* patients who are non-Dutch speaking or understand too little Dutch to fill out the questionnaires

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5200 (Estimated)
Dates: Start 2005-10; Primary Completion 2009-02 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Extent of guideline adherence after approximately one year (measured by a specific set of guideline-derived indicators, formulated beforehand by the research group) | half year after intervention
Costs of both Implementation strategies | half year after intervention

SECONDARY OUTCOMES:
Psychosocial patient characteristics after one year: fear, depression, satisfaction | half year after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rosella PMG Hermens, MSc, PhD, Principal Investigator — Centre for Quality of Care Research; Jan AM Kremer, MD, PhD, Principal Investigator — Department of Obstetrics and Gynecology, Radboud University Nijmegen Medical Centre; Didi D Braat, Prof. MD PhD, Study Chair — Department of Obstetrics and Gynecology, Radboud University Nijmegen Medical Centre; Richard PT Grol, Prof. PhD, Study Chair — Centre for Quality of Care Research; E Adang, Study Director — Department of Medical Technology Assessment, Radboud University Nijmegen Medical Centre; J MM van Lith, MD, PhD, Study Director — Dutch Society of Obstetrics and Gynecology; G Zielhuis, Prof PhD, Study Director — Department of Epidemiology and Biostatistics, Radboud University Nijmegen Medical Centre
Locations (16):
- Netherlands (16):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Gelre Ziekenhuizen, Apeldoorn
  - Rijnstate Ziekenhuis, Arnhem
  - Maasziekenhuis Pantein, Boxmeer
  - ZBC stichting Geertgen, De Mortel
  - Slingeland Ziekenhuis, Doetinchem
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - st Antonius Ziekenhuis, Nieuwegein
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Bernhoven Ziekenhuis, Oss
  - Rivierenland Ziekenhuis, Tiel
  - Bernhoven Ziekenhuis, Veghel
  - Maxima Medisch Centrum, Veldhoven
  - Streekziekenhuis Zevenaar, Zevenaar

REFERENCES:
- [Derived] Mourad SM, Hermens RP, Liefers J, Akkermans RP, Zielhuis GA, Adang E, Grol RP, Nelen WL, Kremer JA. A multi-faceted strategy to improve the use of national fertility guidelines; a cluster-randomized controlled trial. Hum Reprod. 2011 Apr;26(4):817-26. doi: 10.1093/humrep/deq299. Epub 2010 Dec 6. PMID 21134950
- See also: website of the Centre for Quality of Care (WOK) — http://www.wokresearch.nl